CLINICAL TRIAL: NCT03206489
Title: Nasal High Frequency Oscillation for Respiratory Distress Syndrome in Preterm Twins Infants
Brief Title: Nasal High Frequency Oscillation for Respiratory Distress Syndrome in Twins Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Principal Investigator, Ma Juan, director, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: twins with HFO
Record Dates: First submitted 2017-06-26; First posted 2017-07-02 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Nasal High Frequency Oscillation Ventilation
MeSH Terms: interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Intervention Model Description: noninvasive high-frequency ventilation (nHFOV) and nasal continuous positive airway pressure (nCPAP) are used as primary mode of ventilation in preterm twins infants with RDS
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nHFOV (Experimental): noninvasive high-frequency ventilation (nHFOV) is used as a primary mode of ventilation in one of the preterm infants with respiratory distress syndrome
  Interventions: Device: noninvasive high-frequency ventilation (nHFOV)
- nCPAP (Active Comparator): nasal continuous positive airway pressure (nCPAP) is used as a primary mode of ventilation in another of the preterm infants with respiratory distress syndrome
  Interventions: Device: nasal continuous positive airway pressure (nCPAP)

INTERVENTIONS:
Device: noninvasive high-frequency ventilation (nHFOV) — noninvasive high-frequency ventilation (nHFOV) as a primary mode of ventilation in one of the preterm twins infants with respiratory distress syndrome
  Arms: nHFOV
Device: nasal continuous positive airway pressure (nCPAP) — nasal continuous positive airway pressure (nCPAP) as a primary mode of ventilation in another of the preterm twins infants with respiratory distress syndrome
  Arms: nCPAP

SUMMARY:
The investigators compared advantages and disadvantages of two forms of noninvasive respiratory support -noninvasive high-frequency oscillatory ventilation (nHFOV) or nasal continuous positive airway pressure (nCPAP) -as a primary mode of ventilation in preterm twins infants with respiratory distress syndrome

DETAILED DESCRIPTION:
Invasive ventilation is related to development of adverse pulmonary and nonpulmonary outcomes in ventilated infants. Various modes of noninvasive respiratory support are being increasingly used to minimize the incidence of bronchopulmonary dysplasia (BPD). The aim of this trial to compare the effects of noninvasive high frequency oscillatory ventilation (NHFOV) and nasal continuous positive airway pressure (NCPAP) in preterm twins infants as the primary mode.

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age (GA) is from 26 to 37 weeks;
2. Diagnosis of respiratory distress syndrome. The diagnosis of respiratory distress syndrome will be based on clinical manifestations (tachypnea, nasal flaring and or grunting) and chest X-ray findings;
3. Respiratory distress syndrome Silverman score >5;
4. Informed parental consent has been obtained.

Exclusion Criteria:

1. Severe respiratory distress syndrome requiring early intubation according to the American Academy of Pediatrics guidelines for neonatal resuscitation7;
2. Major congenital malformations or complex congenital heart disease;
3. Group B hemolytic streptococcus pneumonia, septicemia, pneumothorax, pulmonary hemorrhage;
4. Cardiopulmonary arrest needing prolonged resuscitation;
5. transferred out of the neonatal intensive care unit without treatment.

Ages: 30 Minutes to 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
intubation | during the first 7 days after birth
  the baby is re-intubated.

SECONDARY OUTCOMES:
Bronchopulmonary dysplasia(BPD) | at a post-menstrual age of 36 weeks or at discharge
  BPD was defined according to the National Institutes of Health consensus definition
Bayley Scales of Infant Development | 30 months after birth
  scores of Bayley Scales of Infant Development at 2 months old and 2 years old

CONTACTS AND LOCATIONS:
Overall Officials: Shi Yuan, PhD,MD, Study Director — Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Locations (1):
- Daping Hospital and the Research Institute of Surgery of the Third Military Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No